CLINICAL TRIAL: NCT05166382
Title: Impact of SomaSignal Tests on the Choice of Glucose-lowering Medications: An Adaptive Implementation Study
Brief Title: Impact of SomaSignal Tests on the Choice of Glucose-lowering Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: SomaLogic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21-4510
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
Keywords: Proteomics; T2D; Type 2 diabetes mellitus; CVD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Providers will be randomized into informed vs uninformed groups. The randomization will occur at each clinic individually to assure equal distribution of informed vs uninformed providers in each clinic. Patients will be assigned a group based on their providers randomization.
Who Masked: Participant, Care Provider
Masking Description: Providers and participants in the uninformed arm will not receive CVD-T2D test results until the second research visit in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: SomaSignal Informed Medical Management (CVDT2D test, informed) (Experimental): Blood draw for cardiovascular CVDT2D test at baseline and 6 months (+/- 30 days). SomaSignal Test results will be sent to the providers and then shared with study participants. Participants' medical record will be reviewed, and they may be contacted within 30 days after baseline and 6-month visits to review changes in treatment strategy (nothing, add/remove medication, etc.) made at visit.
  Interventions: Behavioral: Informed of results from SomaSignal Cardiovascular Risk Test in Type 2 Diabetes (CVD-T2D)
- Group 2: Standard of Care (CVDT2D test, uninformed) (Placebo Comparator): Similar to group 1 but SomaSignal CV test results will not be provided to participants until after the intervention period.
  Interventions: Behavioral: Not informed of results from SomaSignal Cardiovascular Risk Test in Type 2 Diabetes (CVD-T2D)

INTERVENTIONS:
Behavioral: Informed of results from SomaSignal Cardiovascular Risk Test in Type 2 Diabetes (CVD-T2D) — Providers and patients will be informed of CVD-T2D test results that predict the risk of cardiovascular events over the next 4 years after their first research visit.
  Other Names: Informed
  Arms: Group 1: SomaSignal Informed Medical Management (CVDT2D test, informed)
Behavioral: Not informed of results from SomaSignal Cardiovascular Risk Test in Type 2 Diabetes (CVD-T2D) — Providers and patients will be informed of CVD-T2D test results that predict the risk of cardiovascular events over the next 4 years after their second research visit.
  Other Names: Uninformed
  Arms: Group 2: Standard of Care (CVDT2D test, uninformed)

SUMMARY:
The purpose of this study is to learn more about using a proteomic test called the SomaSignal Cardiovascular (CV) Risk Test in Type 2 Diabetes (CVD-T2D) to improve medical care for patients.

ELIGIBILITY:
Inclusion Criteria: Provider

* Licensed provider actively practicing medicine at a UC Health clinic that routinely provides medical treatment for patients with type 2 diabetes

Inclusion Criteria: Patient

* Patients receiving care at a UC Health system
* Age 40 years or older
* Type 2 Diabetes
* Eligible for (per drug label/guidelines) at least one of the following classes: SGLT2i, PCSK9i, GLP-1 RA
* Able to provide consent

Exclusion Criteria:

* Use of SGLT2i , GLP1RA and PCSK9i within the 3 months prior to enrollment
* Systemic Lupus Erythematous (SLE)*
* Pregnancy (as determined by self report)
* Intolerance or contraindication for use of both GLP1RA and SGLT2i
* History of, an active, or untreated malignancy, in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years prior to, or are receiving or planning to receive therapy for cancer, at screening

  * Samples provided by patients with SLE may fail to produce results or may produce inaccurate results because autoantibodies in the patient plasma may interact with the DNA-based reagents used in the assay

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Prescription rates of cardioprotective medications in the informed group vs uniformed group at Baseline | Baseline
  Determine whether risk stratification results from SomaLogic's CVDT2D test leads to risk concordant changes in prescriptions and/or medical management through a patient and provider completed questionnaire. Questionnaire is a binary measurement of "prescribed medicine?" with possible answers "Yes" or "No". Number of participants prescribed medication will be reported.
Prescription rates of cardioprotective medications in the informed group vs uniformed group at Month 6 | 6 months
  Determine whether risk stratification results from SomaLogic's CVDT2D test leads to risk concordant changes in prescriptions and/or medical management through a patient and provider completed questionnaire. Questionnaire is a binary measurement of "prescribed medicine?" with possible answers "Yes" or "No". Number of participants prescribed medication will be reported.

SECONDARY OUTCOMES:
Change in protein predicted risk: SomaLogic CVDT2D test | Baseline, 6 months
  Longitudinal changes in protein-predicted risk as measured by SomaLogic CVDT2D test over 6 months
Change in protein predicted risk: biomarkers | Baseline, 6 months
  Longitudinal changes in protein-predicted risk as measured by conventional biomarkers of risk over 6 months
Standard of care risk assessment: body mass index (BMI) at baseline | Baseline
  Body mass index (BMI) measures a person's weight in kilograms divided by the square of the person's height in meters. Scores between 18.5 and 24.9 indicate a healthy weight.
Standard of care risk assessment: body mass index (BMI) at 6 months | 6 months
  Body mass index (BMI) measures a person's weight in kilograms divided by the square of the person's height in meters. Scores between 18.5 and 24.9 indicate a healthy weight.
Standard of care risk assessment: Atherosclerotic Cardiovascular Disease risk calculator (ASCVD) at baseline | Baseline
  The Atherosclerotic Cardiovascular Disease risk calculator (ASCVD) measures the estimated risk of cardiovascular disease over the next ten years. Possible scores range from <5% to >/=20%, with higher scores indicating a worse outcome.
Standard of care risk assessment: Atherosclerotic Cardiovascular Disease risk calculator (ASCVD) at 6 months | 6 months
  The Atherosclerotic Cardiovascular Disease risk calculator (ASCVD) measures the estimated risk of cardiovascular disease over the next ten years. Possible scores range from <5% to >/=20%, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Neda Rasouli, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Aanchal Gupta, Aurora, Colorado, United States